### Information Sheet for Children and Adolescents (Subjects Ages 7-14)

TITLE: Comparison of Ideal vs. Actual Weight Based Factor Dosing

PROTOCOL NO.: None

WIRB® Protocol #20162706

STUDY00000329

**SPONSOR:** WA State Health Care Authority

**CO-INVESTIGATORS:** Rebecca Kruse-Jarres, MD, MPH

921 Terry Avenue

Seattle, Washington 98104

**United States** 

Amanda Blair, MD

MB.8.501 - Hematology-Oncology

4800 Sand Point Way NE Seattle, Washington 98105

**United States** 

SITE(S): Washington Center for Bleeding Disorders at Bloodworks

Northwest 921 Terry Ave

Seattle, Washington 98104

**United States** 

Seattle Children's Hospital 4800 Sand Point Way NE Seattle, Washington 98105

**United States** 

Seattle Children's 1900 9<sup>th</sup> Avenue

Seattle, Washington 98101

**United States** 

STUDY RELATED

**PHONE NUMBER(S):** Rebecca Kruse-Jarres MD, MPH

206-689-6507

206-292-6525 option # 3 (24 hours) and (ask for the Hemophilia

physician on call)

Amanda Blair 206-987-2106

STUDY-

**COORDINATOR(S):** Heidi Thielmann, PhD

206-689-6234

Kimberly Starr 206-884-8163

#### Why should I be in the study?

We are doing a research study. We want to learn more about the factor products you take for your hemophilia.

#### What do I have to do?

You can say yes and join this study. Your doctor would like to collect some information about your health from your medical record in order to see if you will qualify for this study. Your doctor or nurse might ask you a few questions about your health. You do not have to answer any question you do not want to. If you join the study, you will come to the clinic twice to have a factor dose. Then you will have your blood taken at different times on different days after your factor dose.

#### Will it hurt?

It will feel like a pinch when you give blood. It will hurt for a minute. Sometimes the place where the needle went in can be sore for a while or you might have a bruise for a few days.

#### How will it help?

This study will not help you. The things we learn from this study might help people with hemophilia.

APPROVED AS MODIFIED Aug 07, 2017 WIRB®

# Do I have to be in this study?

Your mother/father said it would be ok for you to participate in this research project. If you do not want to be a part of this research project, you will still get the same care that you have been getting. If you don't want to be in this study, that is okay. You can change your mind later if you want to stop.

## Can I ask questions?

You may ask us any questions now that you want. If you think of a question later on, you can ask your parent. Your parent can call us to ask a question too.